CLINICAL TRIAL: NCT00390949
Title: Impact and Process Evaluation of Integrated Community and Clinic-based HIV-1 Control: a Cluster-randomised Trial in Eastern Zimbabwe
Brief Title: Scientific Evaluation of Peer Education and STD Treatment to Reduce the Spread of HIV in Zimbabwe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Biomedical Research and Training Institute (Other)
Responsible Party: Principal Investigator, Simon Gregson, Professor of Demography and Behavioural Science, Imperial College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PC3239_DFID
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Results first posted 2019-08-29 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: HIV Infections
Keywords: HIV prevention; Zimbabwe; Core groups; Peer education; Syndromic management; Commercial sex workers; Condom distribution; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

ARMS (2):
- Intervention arm (Experimental): Peer education with female sex workers and potential male clients. Strengthened syndromic management of STIs with community-based promotion activities
  Interventions: Behavioral: Peer education among commercial sex workers and clients; Behavioral: Condom distribution and promotion; Procedure: Syndromic treatment of sexually transmitted infections; Procedure: Systemic counselling for STI patients
- Control (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Peer education among commercial sex workers and clients
  Arms: Intervention arm
Behavioral: Condom distribution and promotion
  Arms: Intervention arm
Procedure: Syndromic treatment of sexually transmitted infections
  Arms: Intervention arm
Procedure: Systemic counselling for STI patients
  Arms: Intervention arm

SUMMARY:
The purpose of this study is to determine whether community-based peer education and condom distribution combined with improved treatment of sexually transmitted infections are effective in reducing the spread of HIV infection in a sub-Saharan African population

DETAILED DESCRIPTION:
Background and Literature Review

The Spread and Early Demographic Impact of HIV in Zimbabwe

High levels of HIV prevalence and incidence have been recorded in Zimbabwe since sentinel surveillance was introduced in 1990. Prevalence levels in excess of 40% have been recorded among women attending antenatal clinics in a number of urban centres [1,2]. In a cohort study of male factory workers conducted in Harare between 1993 and 1995, 19% of participants were found to have the infection at enrolment and an incidence rate of 2.93% per annum was recorded [3]. However, rural areas - where 70% of the country's population are based - are experiencing some of the highest rates of incidence at the current time. In Mberengwa, Midland Province, HIV prevalence among pregnant women increased from under 8% in 1992 to 25% in 1994 [4].

In a study in two rural areas of Manicaland Province, we also found high levels of HIV infection at antenatal clinics in 1993-94 - 24% and 14%, at the growth points in the Honde Valley and the Rusitu Valley, respectively. Further data from the Honde Valley in 1996 indicate that incidence remains high (2-4%). Significant increases in adult and infant mortality and in orphanhood were recorded. The cause-specific and age-patterns of increase indicate that these are due primarily to HIV infections. Sexual intercourse with casual partners is common and condom use is low. In qualitative studies, high proportions of men, but relatively few women, reported recent casual partnerships. Mathematical model simulations indicate that this pattern of behaviour could explain the greater excess mortality that was recorded among males, given a recent - last 4-5 years - escalation of the HIV epidemic in rural areas. Other ulcerative and non-ulcerative sexually transmitted diseases (STDs) are common, but only 2% of respondents were aware that STDs can facilitate HIV transmission [5 8].

Mathematical model projections, based on our understanding of the predominant behaviour pattern and fitted to observed trends in HIV prevalence, also indicate that further increases in adult and early childhood mortality are to be expected. Results from these simulations and empirical findings from Uganda suggest that these increases will result in adverse indirect effects, including high proportions of children experiencing orphanhood and distortions in the age- and sex-distribution of the population [9,10]. These effects may be compounded by fertility change. Birth rates are declining in rural areas of Zimbabwe at present and the HIV epidemic may re-enforce this decline through changes in behaviour or underlying fecundity [11]. Women with HIV infection are reported as having lower fertility than other women in Ugandan studies [12] and results from our research in Manicaland indicate that behaviour changes which would tend to re-enforce the existing decline in birth rates may be beginning to occur [7].

HIV Prevention Strategies

Mathematical model simulations have demonstrated the potential for reducing the incidence of new HIV infections through biomedical and behavioural interventions. The benefits of early interventions and of targeting interventions at core groups have been emphasized [13,14]. Targeted interventions are liable to be less effective if introduced after high levels of HIV prevalence have been reached. Their success will also depend on the level of heterogeneity in sexual activity which exists within a population and the predominant pattern of mixing between different risk groups [15]. Combinations of intervention approaches can act additively and even synergistically [16].

In one set of simulations, based on epidemiological data from rural Uganda, it was demonstrated that a combined biomedical and behavioural intervention which (a) increased condom use in contacts between men and casual sex partners to 50%, (b) reduced the frequency of these contacts by 50%, and (c) reduced the average duration of STD episodes by 50%, could reduce HIV incidence by 50% in the first year and 80% over ten years. Empirical studies have shown that changes of this nature are possible and can lead to large reductions in HIV incidence. In Nairobi, health education and condom promotion led to an increase in condom use among commercial sex workers from 8% to 66%. Condom use was associated with a 3-fold reduction in risk of sero-conversion [17]. In Zimbabwe, large-scale condom promotion programmes were associated with 48% and 53% reductions in STD cases over three years, in Bulawayo and Mutare, respectively. Most of these reductions were achieved within the first year of the intervention [18]. In a study of 752 male factory workers in Mwanza, Tanzania, counselling at an STD clinic contributed to significant reductions in reported high-risk behaviour - eg: the proportion with more than one sexual partner in the preceding month fell from 22% to 12% - and a large (63%) - but non-significant - reduction in HIV incidence [19,20]. In a randomized control trial in rural areas around Mwanza, improved diagnosis and treatment of STDs was associated with a 42% reduction in the incidence of new HIV infections over a two-year period [21,22].

While these examples demonstrate the effectiveness of individual interventions, there remain shortages of scientific evaluations of combined approaches and of programmes which are sustainable within rural communities, where the majority of sub-Saharan African populations are based and where HIV is now spreading rapidly [23]. Studies of this kind are essential to establish the effectiveness of different intervention strategies and to provide demonstration models which can be used to promote the implementation of interventions which are appropriate and cost-effective.

Care and Support Interventions

As HIV epidemics begin to cause higher morbidity, mortality, orphanhood and socio-economic hardship, affected communities require interventions which provide support in coping with these problems, particularly so, as institution-based solutions become less viable. This need is often upper-most in people's minds, so that prevention programmes which are linked to care initiatives - especially where infected community members are supported and involved in prevention - are considered likely to be most effective [24]. Few systematic evaluations have been conducted to assess the effectiveness of existing care and support models. However, it is clear that programmes which include a high level of external biomedical input are unlikely to be financially sustainable [25]. On the other hand, early evaluations indicate that initiatives which encourage local community ownership and participation, whilst more limited in scope, can be extremely cost-effective [26].

Community-Based, HIV Prevention, Care and Support Intervention Strategy for Rural Zimbabwe

In the light of the above, it is proposed to initiate a community-based, combined HIV prevention, care and support intervention in the Honde Valley and neighbouring areas of the Mutasa District of rural Manicaland. The proposed intervention will ultimately cover an area of approximately 2,750 square kilometres, comprising a population of around 170,000 people. The project will be a collaborative programme promoted by Family AIDS Caring Trust (FACT) and the Biomedical Research and Training Institute (BRTI) and involving local community and church groups and local Ministry of Health personnel. FACT is a Zimbabwean NGO based in Mutare, the provincial capital of Manicaland, and has a well-deserved reputation as an organization which has pioneered innovative community-based HIV control activities in Zimbabwe. Its' established projects include prevention and support programmes in both urban and rural areas of the province. FACT will be responsible for behavioural (including condom promotion and distribution activities and community-based promotion of STD services), support and care aspects of the programme. BRTI is a relatively recently-formed organization based in Harare with strong links with the University of Zimbabwe Medical School, the Blair Research Institute and other parts of the Ministry of Health and Child Welfare. BRTI has considerable expertise in STD diagnostic methods and treatment regimes and would be responsible for this aspect of the intervention and evaluation, in close co-operation with the Ministry of Health in Manicaland. It serves a similar function in established HIV control programmes elsewhere in Zimbabwe. BRTI would also act as employer for staff engaged to carry out the fieldwork for the intervention evaluation.

PLAN International have recently extended their area of operation in Zimbabwe to include the Honde Valley and have agreed to provide funding for the HIV intervention programme for a minimum period of four years. PLAN maintain routine records on a number of key impact indicators so that the projects they sponsor can be assessed. It may be possible to develop these systems so that they provide information on indicators of the impact of the HIV epidemic and the effectiveness of AIDS control activities - eg: programme coverage and success in targeting - which could be used in this study and for long-term monitoring purposes.

The proposed intervention strategy appears to have good potential for sustainability and replication. Factors which support this view include the emphasis on local community involvement, the low cost of external inputs, the well-established local NGO partner, Ministry of Health support, and the presence of a rural-based, community-orientated funding organization with a substantial international funding base and a long-term commitment to extending the scope of its activities in Zimbabwe. Descriptions of the principal intervention elements are contained in separate documents attached to this proposal.

Objectives of the Study

The principal objectives of the study are as follows:

1. To scientifically evaluate the impact and cost-effectiveness of a combined behavioural and STD-control intervention strategy to slow the spread of HIV infections in rural Zimbabwe; and
2. To extend recent monitoring of the demographic impact of the HIV epidemic in a rural area of Zimbabwe.

Subsidiary aims include validation of innovative methods for data collection on HIV, other STDs - ie: using saliva samples [35] - and sexual behaviour in rural settings (all subject to final pre-test in the pilot study) and for estimating HIV incidence from cross-sectional prevalence data [27]; evaluation of antenatal clinic data as a source of information on HIV levels within the general population; and development of methods for routine evaluation of community-owned support programmes for individuals and families affected by heightened experience of chronic morbidity and mortality.

Methodology

Experimental Design for the Intervention Trial

Six pairs of sub-communities (clusters), matched for similar levels of key factors affecting the spread of HIV, will be identified in the vicinity of the Honde Valley. Four of these pairs are likely to be within commercial estates - tea, coffee, forestry and orchards - and two in communal farming areas. Each sub-community will be chosen so that it includes a health clinic where improved STD services can be made available. The behaviour and STD-control intervention will be introduced in one cluster within each pair on a phased basis over a period of twelve months - ie: one new cluster every two months. In each case, a baseline survey for the evaluation will be conducted in the intervention and comparison clusters in the two-month period immediately prior to the introduction of the programme. For the evaluation, 1,000 respondents will be enrolled within a sector of each sub-community following an initial household census - half of those enrolled will be men aged 17-49 years and half will be women aged 15-39 years. Individuals who usually reside in the household will be eligible for full participation in the study - i.e.: recruitment will be on a de jure basis - in order to increase follow-up and reduce within-group heterogeneity. Within a household, the random selection process used will avoid instances where a husband and wife or more than one wife are enrolled and thereby reduce correlation of outcomes within individual clusters. Respondents in each pair of clusters will be surveyed again two years months after the baseline visit. Records will be kept on an anonymous basis but a mechanism will be put in place to enable the data to be linked within and between survey rounds.

Outcome indicators will include knowledge about HIV and AIDS, sexual behaviour indicators - partner acquisition and partnership duration, mixing patterns and condom use - incidence of HIV and selected STD infections, and health-seeking behaviour indicators. Sample sizes were calculated to give an 80% power at the 95% significance level, comparing the matched intervention and comparison clusters, for a range of different outcome variables. The formulae used in these calculations take account of possible between-cluster and - in the case of prevalence - within-cluster variability [22,28]. Given the level of spatial mobility which exists within the Honde Valley area, some diffusion effect is likely to be present. This has been reflected in the sample size computations through the use of conservative anticipated excess reductions in the intervention clusters. We estimate that a sample size of 1,000 individuals per cluster will yield a minimum of 700 observations, after accounting for loss to follow-up. In the case of the HIV incidence calculations, these observations will provide 1,120 susceptible person-years of observation, after allowing for a baseline prevalence in the general adult population of 20%. Under these conditions, an initial sample size of 1,000 per cluster should be sufficient to permit detection of a 40% excess reduction in HIV incidence, given a baseline annual incidence of 2% or higher. This sample size should also enable us to detect, inter alia, a 40% lower incidence of new HSV2 and trichomoniasis cases among individuals not infected at baseline and a 40% reduction in reported casual relationships without the use of condoms, given a baseline prevalence of 10% or over. Evidence from model simulations and empirical studies suggests that the excess reduction in HIV incidence required is plausible given a combined intervention strategy [19,29]. Furthermore, the required excess reductions in STDs and high-risk behaviour should be attainable. Reductions in these factors, of the order indicated, would, if demonstrated, represent strong indirect evidence that the intervention strategy is slowing the spread of HIV infections. Reduction in other STDs would be a significant benefit, in itself, given the morbidity and adverse fertility consequences they frequently cause.

Data Collection: Quantitative and Qualitative Methods

Quantitative data will be collected on the intervention trial outcome measures summarized above, principally through the two-round survey. A cohort of participants for this survey will be recruited in a household census within each of the twelve study areas. The second round of the study will be conducted two years after the first visit in each area and will involve a repeat household census and further detailed interviews with the original participants. The population-based survey will also provide data on process indicators, including measures of contact with the intervention programme - eg: numbers of meetings attended and visits received from programme personnel - and utilization of programme services - eg: free condoms, revolving loans, care support, STD diagnosis and treatment - and other potential determinants of key outcomes, including socio-economic and demographic factors, and personal experience of HIV-related morbidity and mortality. Data will be collected on demographic indicators - eg: age- and gender-specific mortality, recent fertility, orphanhood and household composition - in the household and individual interviews, using standard demographic methods [30,31]. Quantitative data will also be collected on HIV prevalence at antenatal clinics, so that the representativeness of data from this source can be evaluated. Qualitative data on sexual and health-seeking behaviour and obstacles to behaviour change will be collected in focus-group discussions, pocket-chart voting sessions and key-informant interviews [32,33] and employed to aid questionnaire design and validation and in interpretation of statistical results. These methods were used successfully in our previous study [7]. However, to strengthen this aspect of the current proposal, additional input on the design and implementation of appropriate ethnographic methods will be received from a collaborator from the LSE (Dr. Campbell).

Steps will be taken to develop the good working relationship already formed with the Honde Valley community, to mobilize community support for the research and provide reassurance that information given will be treated as strictly confidential. Thus, we hope to achieve high participation and follow-up rates and more reliable information. Preliminary meetings will be held with community leaders to explain the purpose of the study and the research procedures. Similar information will be given to each prospective participant prior to their decision on enrolment. Data collection methods such as self-completion questionnaires - 96% and 45% of women aged under 50 years, living in the Honde Valley, have received primary and secondary education, respectively, and literacy levels among men are higher than those for women [7] - and secret balloting, which avoid the need for participants to reveal personal information to enumerators directly and thus reduce under-reporting of sensitive information [34], have been field-tested and will be pre-tested further in the pilot study and used where feasible. Similarly, the possibility of using less invasive media such as saliva, urine or blood spot samples for HIV and STD testing is being investigated with the Public Health Laboratory in Harare [35]. The reliability and acceptability of these methods as applied in rural settings will also be field-tested in the pilot study.

Questionnaires will be translated into the local Manyika dialect of Shona, back-translated and pre-tested in the pilot study. Data entry and validation will be undertaken using SPSS-PC+. Appropriate data entry forms will be designed for each section of the survey questionnaires and skip-rules, range checks etc will be employed to reduce data entry errors. BRTI/Blair staff have considerable experience of using SPSS-PC+ for data entry.

Data Analysis: Scope and Methods

Reliability and validity checks will be conducted to assess the quality of the quantitative data [36]. Data analysis will be conducted using statistical software - eg: STATA and SAS - and mathematical models of HIV incidence, which are based on underlying biomedical, behavioural and demographic determinants of HIV infections [37,38]. Statistical analyses will include tests for the significance of differences arising between paired intervention and control clusters [39,40] and tests for impact of contacts with the intervention programme and other possible determinants on changes in reported behaviour. The impact of the HIV epidemic on mortality will be monitored using longitudinal survey data and official vital registration records. Impact on fertility will be assessed by comparing birth rates among infected and uninfected individuals, controlling for other key determinants including age, education, religion and history of STDs. Crude birth rates, crude death rates and levels of natural population increase will be estimated from the survey data and the trends evaluated [12]. Coverage and impact of care/support interventions will be investigated. HIV prevalence estimated from the population-based survey will be compared with estimates from women attending antenatal clinics to assess the representativeness of the latter. Adjustments will be made in data analysis for the matched-pair design of the study. Data from the study will be used to evaluate new methods for estimating incidence from cross-sectional HIV prevalence surveys [27].

Ethical Considerations

Informed consent will be sought as a condition for enrolment in the study. This will be in written form wherever literacy levels allow - which is expected to be in the great majority of cases. A written statement in the local dialect of shona will be provided explaining the purpose of the study and all aspects, benefits and risks of participation. The statement will make it clear that participants have the right to withdraw from the study at any time. Time will be allowed for prospective participants to read the statement, to ask questions and consider their decision. The statement will be read aloud to prospective participants who are unable to read themselves. Enumerators will be trained to do this in a balanced manner so as to avoid possible coercion.

Participants will be given the opportunity to receive HIV-1 test results. Preliminary counselling will be offered during study interviews. Where participants indicate that they would like to be advised as to their own HIV-1 serostatus, appointments will be arranged for them to visit a local clinic where a free counselling and testing service will be made available. Standard Ministry of Health and Child Welfare and WHO procedures will be followed throughout, with further serological tests being undertaken as required.

Participants who test positive for other sexually transmitted diseases will be advised of their results and a free treatment service will be offered wherever possible (eg: for trichomoniasis). Less invasive media such as urine and saliva will be used for the collection of samples for HIV-1 and STD testing. Where blood samples are sought, blood spots rather than venipuncture will be used. Appropriately qualified and trained personnel will be employed to collect the samples.

Rigorous procedures will be maintained throughout the study to ensure full confidentiality of information obtained from participants. Data protection and anonymization procedures will be implemented and computerized matching methods will be used to ensure that access to linked data will be strictly limited to the principal investigators only, with the single exception that appropriate medical staff will be given access to results of HIV-1 or STD tests where participants wish to be informed of their results or to be offered treatment. The procedures will be such that staff, study participants and other individuals are not able to deduce individual HIV-1, STD and sexual behaviour details by applying exclusion and inclusion criteria. Confidential voting methods will be employed in the collection of sexual behaviour information so as to avoid the need for participants to impart personal information to enumerators.

Benefits to participants will include participation in prevention, care and support activities in the intervention areas (see separate description of intervention activities). Subject to confirmation that these activities are effective, the researchers and programme managers are committed to ensuring that similar programmes will be introduced within each control area two years after the study is initiated in that area. In all areas, participants will be offered free treatment of STDs identified in the survey. Free information sheets on HIV-1 infection and AIDS which address gaps in information identified in the earlier study in Honde Valley will be made available to study participants in all areas during the baseline survey. Risks of participation in the research team or as a community member are believed to be low. Rigorous procedures are to be followed to avoid needle-stick injuries and to ensure confidentiality of information obtained, standard treatments will be offered for STDs diagnosed and established tests and associated procedures, which have proved to be very reliable in Zimbabwean settings, will be used for HIV-1 diagnosis, in particular, where results are to be made available to participants.

Dissemination of study results will be done through the Biomedical Research and Training Institute (BRTI) and Blair Research Institute with approval from the Ministry of Health and Child Welfare. An original copy of the data set from the study will remain in Zimbabwe at BRTI and/or Blair. Approval for the study will also be obtained from the Central Oxford Research Ethics Committee in the United Kingdom prior to implementation.

Personnel, Workplan and Location of Project Activities

Dr. Gregson will manage and co-ordinate the proposed research project with expert epidemiological and statistical support from the Blair Research Institute in Harare and the Wellcome Trust Centre for the Epidemiology of Infectious Disease, at Oxford University (Dr. Chandiwana, Professor Anderson, Dr. Garnett and Dr. Donnelly), social psychology and ethnographic support from BRTI, the London School of Economics and the University of Natal (Mr. Tom Zhuwau, Dr. Cathy Campbell, Professor Eleanor Preston-Whyte and Professor Linda Richter), and biomedical support from BRTI (Professor Mason and Mr. Ocean Tobaiwa). Within the team we have considerable management and administrative as well as research experience and in a previous project we demonstrated the ability to develop and conduct a successful fieldwork-based scientific research project, given the level of technical and logistical support envisaged in this proposal. Zimbabwe has a good supply of well-qualified personnel in most disciplines and staff with appropriate sociological, demographic and/or medical expertise will be recruited. All staff will be given in-depth training in the specific requirements of the study. A summary schedule of project activities over time is attached.

Intended Use of Results

The results will be disseminated through seminars, workshops and publications in local and international journals. In these ways, we will seek to promote greater awareness of the level of effectiveness of the intervention strategy evaluated in the given context.

ELIGIBILITY:
Inclusion criteria:

Age: Males aged 17-54 years; females aged 15-44 years at last birthday Residence: Slept in a household in the study areas on at least 4 nights in the last 30 days

Exclusion criteria:

Age: Males below the age of 17 years at last birthday or aged 55 years or above; females below the age of 15 years at last birthday or aged 45 years or above Residence: Did not sleep in a household in the study areas on at least 4 nights in the last 30 days

Ages: 15 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 9454 (Actual)
Dates: Start 1998-07 (Actual); Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Gregson, DPhil, Principal Investigator — Imperial College London; Stephen Chandiwana, PhD, Principal Investigator — Biomedical Research and Training Institute
Locations (1):
- Biomedical Research and Training Institute, Harare, Zimbabwe

REFERENCES:
- [Background] Campbell C, Scott K, Mupambireyi Z, Nhamo M, Nyamukapa C, Skovdal M, Gregson S. Community resistance to a peer education programme in Zimbabwe. BMC Health Serv Res. 2014 Nov 19;14:574. doi: 10.1186/s12913-014-0574-5. PMID 25407818
- [Result] Gregson S, Garnett GP, Nyamukapa CA, Hallett TB, Lewis JJ, Mason PR, Chandiwana SK, Anderson RM. HIV decline associated with behavior change in eastern Zimbabwe. Science. 2006 Feb 3;311(5761):664-6. doi: 10.1126/science.1121054. PMID 16456081
- See also: Manicaland HIV/STD Prevention Project website — http://www.manicaland-project.org/
- See also: Biomedical Research and Training Institute, Harare — http://www.brti.co.zw/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from six pairs of sub-communities matched on socio-economic criteria
Groups:
- Control Arm: Control communities were to receive standard Government services including basic syndromic STI management, condom distribution from health clinics and Zimbabwe National Family Planning Council outlets, homebased care, and limited HIV/AIDS-focussed IEC activities (e.g., occasional AIDS-awareness meetings and distribution of posters and leaflets). In addition, social marketing of male and female condoms would be provided through an ongoing national programme.
- Intervention Arm: In addition to the standard-of-care services provided in the control arm, the intervention communities were to receive targeted and population-level activities to promote safer sexual behaviour and to improve treatment of STIs that facilitate HIV-1 transmission. The intervention strategies were to be implemented by two local nongovernmental organisations and the Zimbabwe Ministry of Health and Child Welfare through an integrated programme of community- and clinic-based activities. The programme design comprised three key components: (1) peer education and condom distribution amongst commercial sex workers and male clients at workplaces and in the general community, supported by income-generating projects; (2) strengthened syndromic management of STI services at local health centres; and (3) open days with HIV/AIDS IEC activities at health centres to promote safer sexual behaviour and to increase the uptake of local STI treatment services.
Period: Overall Study
Arm/Group | Control Arm | Intervention Arm
Started | 4662 | 4792
Completed | 2564 | 2664
Not Completed | 2098 | 2128

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Intervention Arm | Total
Number analyzed (Participants) | 4662 | 4792 | 9454
Age, Customized [Count of Participants; unit: Participants]
  Age group in years: Under 20 | 1138 | 1127 | 2265
  Age group in years: 20-24 | 1036 | 1095 | 2131
  Age group in years: 25-34 | 1338 | 1363 | 2701
  Age group in years: 35-44 | 955 | 1037 | 1992
  Age group in years: 45 and above | 195 | 170 | 365
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2502 | 2632 | 5134
  Male | 2160 | 2160 | 4320
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4662 | 4792 | 9454
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Zimbabwe | 4662 | 4792 | 9454
HIV prevalence [Count of Participants; unit: Participants]
  HIV positive | 999 | 1172 | 2171
  HIV negative | 3663 | 3620 | 7283
More than 5 sexual partners in lifetime [Count of Participants; unit: Participants] | 999 | 1063 | 2062

OUTCOME MEASURES:

1. Primary Outcome: HIV Incidence at the Community Level
Description: Number of new infections occurring per 100 person-years of follow-up
Time Frame: 3 years
Population: General population
Measure: Number (95% Confidence Interval); unit: HIV infections per 100 person-years
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 2564 | 2664
HIV infections per 100 person-years | 1.49 [1.18 to 1.80] | 2.04 [1.68 to 2.40]

2. Secondary Outcome: Self-reported Genital Ulcers
Description: Percentage of sexually-experienced adults reporting genital ulcers
Time Frame: 1 year
Population: Men and women who report having started sex
Measure: Number (95% Confidence Interval); unit: Percentage of sexually active adults
Groups:
- Intervention Arm: Peer education with female sex workers and potential male clients. Strengthened syndromic management of STIs with community-based promotion activities
  Peer education among commercial sex workers and clients
  Condom distribution and promotion
  Syndromic treatment of sexually transmitted infections
  Systemic counselling for STI patients
Arm/Group | Intervention Arm | Control
Number analyzed (Participants) | 2523 | 2409
Percentage of sexually active adults | 9.04 [7.95 to 10.22] | 7.47 [6.45 to 8.60]
Statistical Analysis 1: Comparison: Intervention Arm vs Control; Test type: Superiority; p < 0.05, Regression, Logistic — The p-value reported above is not simply a statement of the threshold for significance used in the study. The p-value for this comparison was calculated at the time of the study and was found to be less than 0.5; Adjustments for community pair, age-group and value of variable at baseline

3. Secondary Outcome: Self-reported Urethral or Genital Discharge
Description: Percentage of sexually-experienced adults self-reporting urethral or genital discharge
Time Frame: 1 year
Population: Men and women who report having started sex
Measure: Number (95% Confidence Interval); unit: Percentage of sexually experience adults
Arm/Group | Intervention Arm | Control
Number analyzed (Participants) | 2528 | 2418
Percentage of sexually experience adults | 11.91 [10.67 to 13.23] | 10.50 [9.31 to 11.80]
Statistical Analysis 1: Comparison: Intervention Arm vs Control; Test type: Superiority; p < 0.05, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Adjusted for community pair, age-group and value of variable at baseline

4. Secondary Outcome: Percentage of Participants Reporting Cessation of Sexually Transmitted Infection Symptoms
Description: Self-reported sexually transmitted infection treatment effectiveness based on self-reported cessation of symptoms
Time Frame: 1 year
Population: Men and women who report having started sex and STI symptoms in past year
Measure: Number (95% Confidence Interval); unit: Percentage of sexually experience adults
Arm/Group | Intervention Arm | Control
Number analyzed (Participants) | 278 | 273
Percentage of sexually experience adults | 71.58 [65.89 to 76.81] | 60.44 [54.37 to 66.28]
Statistical Analysis 1: Comparison: Intervention Arm vs Control; Test type: Superiority; p < 0.05, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]

5. Secondary Outcome: Percentage of Participants Reporting More Than One Casual Partner in the Past 3 Years
Description: Percentage of participants in the survey who report more than one casual partner in the past 3 years
Time Frame: 3 years
Population: Men and women who report having started sex
Measure: Number (95% Confidence Interval); unit: Percentage of sexually experience adults
Arm/Group | Intervention Arm | Control
Number analyzed (Participants) | 2447 | 2302
Percentage of sexually experience adults | 14.59 [13.21 to 16.05] | 13.38 [12.01 to 14.84]
Statistical Analysis 1: Comparison: Intervention Arm vs Control; Test type: Superiority; p < 0.05, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Adjusted for community pair, age-group and value at baseline

6. Secondary Outcome: Percentage of Participants Attending a Peer Education or Other Programme Meeting
Description: Percentage of survey participants reporting having attended a peer-education activity or other intervention programme meeting
Time Frame: 3 years
Population: Adults in the general population followed up from baseline
Measure: Number (95% Confidence Interval); unit: Percentage of adults
Arm/Group | Intervention Arm | Control
Number analyzed (Participants) | 2612 | 2486
Percentage of adults | 20.25 [18.73 to 21.85] | 4.75 [3.94 to 5.66]
Statistical Analysis 1: Comparison: Intervention Arm vs Control; Test type: Superiority; p < 0.05, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Adjusted for community pair and age-group

7. Secondary Outcome: Percentage of Participants Scoring 60% or Above on an Index of HIV/AIDS Knowledge
Description: Index calculated based on responses to a set of survey questions on knowledge about how HIV can be transmitted, factors increasing the risk of HIV transmission, signs and symptoms of HIV/AIDS, and the average durations of HIV infection and survival with AIDS at the time of the study (i.e. in the period prior to availability of antiretroviral treatment). Index scores could range between 0% and 100% with higher scores reflecting greater knowledge about HIV and AIDS.
Time Frame: 3 years
Population: Adults in the general population
Measure: Number (95% Confidence Interval); unit: Percentage of adults
Arm/Group | Intervention Arm | Control
Number analyzed (Participants) | 2683 | 2590
Percentage of adults | 51.40 [49.49 to 53.31] | 47.30 [45.36 to 49.24]
Statistical Analysis 1: Comparison: Intervention Arm vs Control; Test type: Superiority; p < 0.05, Regression, Logistic — [p-value comment as in outcome 2, analysis 1]; Adjusted for community pair, age-group and value at baseline

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 years per participant
Arm/Group | Control Arm | Intervention Arm
Serious Adverse Events (participants affected / at risk) | 0/4662 | 0/4792
Other Adverse Events (participants affected / at risk) | 0/4662 | 0/4792

LIMITATIONS AND CAVEATS:
The study was conducted at the peak of a large HIV epidemic during a period of high inflation and the results might not be generalizable to other epidemiological or structural conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes